CLINICAL TRIAL: NCT06709755
Title: A Hybrid Effectiveness-implementation Trial of an Intervention to Reduce Diabetes-specific Emotional Distress in Teenagers
Brief Title: A Hybrid Effectiveness-implementation Trial to Reduce Diabetes Distress in Teenagers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: American Diabetes Association (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-6418
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes distress; adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STePS in Person. This is the STePS intervention provided in an inperson modality (Experimental): The participants will receive the 9-session STePS intervention in person
  Interventions: Behavioral: Supporting Teen Problem Solving
- STePS Virtual. This is the STePS intervention provided in a virtual format (Experimental): The participants will receive the 9-session STePS intervention virtually
  Interventions: Behavioral: Supporting Teen Problem Solving
- Diabetes Education Group (Active Comparator): The Participants will receive diabete education directed toward adolescents matching time, group experience and homework assignments, delivered virtually
  Interventions: Behavioral: Diabetes Education

INTERVENTIONS:
Behavioral: Supporting Teen Problem Solving — STePS is a group-based, teen-focused intervention aimed at reducing diabetes-specific emotional distress and building diabetes resilience. STePS is grounded in both cognitive-behavioral and social problem-solving theories, which recognize the interrelationships among difficult situations, beliefs related to the cause and consequences of those situations, and the emotional and behavioral consequences of those beliefs, and which addresses problem solving strategies that influences ones' adaptive functioning in real-life social settings, distinguishing between problem solving and solution implementation. STePS reduces distress by teaching: 1) emotion regulation, helping teens learn to link beliefs, emotions, and behaviors; to challenge negative thinking by evaluating the accuracy of one's beliefs; and learning new coping skills.2) perspective taking, helping teens learn to identify their own thinking style.
  Arms: STePS Virtual. This is the STePS intervention provided in a virtual format; STePS in Person. This is the STePS intervention provided in an inperson modality
Behavioral: Diabetes Education — Arm Description: The Participants will receive diabetes education directed toward adolescents matching time, group experience and homework assignments, delivered virtually
  Arms: Diabetes Education Group

SUMMARY:
The investigators will assess both effectiveness (primary) and implementation (secondary) outcomes for a distress-reducing intervention, Supporting Teen Problem Solving (STePS). STePS has already undergone an efficacy trial. The current study allows for evaluating the outcomes of STePS by delivering it in real-world settings, using real-world providers. The investigators will train these behavioral health providers who are already embedded in diabetes clinics to use the STePS intervention. The investigators will also compare two approaches to intervention delivery: in-person versus telehealth. The investigators have recruited 6 different study sites across the country, representing diversity in rural vs. urban, public vs private insurance, as well as in ethnic and racial background of the participants. 360 teens will be enrolled and randomized to either STePS or an educational control group on a 1:1:1 basis at each of our 6 study sites: STePS in-person (n=120), STePS telehealth (n=120), or educational control via telehealth (n=120).

All 3 groups will be delivered as 4.5-month interventions, consisting of 9 sessions offered twice per month. Quantitative data (surveys) will be collected for all participants at baseline, immediately post-intervention, and 6 & 12 months post-intervention. Qualitative data will also be collected post-intervention through focus groups.

Aim 1. To test, in 360 teens across 6 clinical sites, the effectiveness of STePS in improving diabetes- specific emotional distress and preventing worsening glycemic control, both immediately post intervention and over time. Hypothesis 1a: STePS will lead to clinically meaningful and statistically significant improvements in diabetes distress. Hypothesis 1b: STePS will prevent the worsening of glycemic control (A1C and Time in Range). These hypotheses are consistent with the efficacy trial and will prove effectiveness when implemented in real- world settings.

Aim 2. To assess the implementation of STePS among key stakeholders (teen participants, interventionists). Recruitment, enrollment, representativeness, feasibility, acceptability, appropriateness, fidelity, and costs will be assessed as well as preferred implementation approaches. Hypothesis 2a. Stakeholders will find few perceived barriers to implementing STePS and many perceived facilitators for adopting it in their clinical settings. Hypothesis 2b. Implementation strategies will be plausible in diabetes clinics across the country.

DETAILED DESCRIPTION:
Diabetes distress among teens is common and associated with poor glycemic control and poor psychosocial outcomes. Diabetes-specific emotional distress (abbreviated DD in this proposal) is emotional distress culminating from living with diabetes and the burden of relentless daily self-management. Teens are at high risk for DD as diabetes self-management behaviors decline, and glycemic control worsens. Only 17% of teens achieve recommended glycemic targets for time-in-range (TIR) of 70-180 mg/dL and hemoglobin A1c <7.0%.7,8 DD is highly prevalent in teenagers (21%-52%) and is associated with suboptimal glycemic control, and an increased risk of future complications, even when controlling for demographic variables such as race and socioeconomic status. DD is a stronger predictor of A1c than depression. In a study of DD trajectories, teens with higher A1cs at baseline were more likely to experience chronically high levels of DD over time. Alarmingly, prospects do not improve as teens transition to adulthood without treatment. The American Diabetes Association's (ADA), the International Association for Pediatric and Adolescent Diabetes (ISPAD), and NIDDK highlight DD as a vital intervention target for youth.

Supporting Teen Problem Solving (STePS) is a highly scalable, group-based DD intervention for teens that builds diabetes resilience. In the sole efficacy trial to date, our team found that STePS demonstrated: 1) continued improvements in DD over time, with effect sizes increasing up to 3 years post-intervention, a statistically significant and clinically meaningful outcome, and 2) prevented worsening A1c, with 3-year post-intervention results of stable A1c. The latter is noteworthy because longitudinal evidence shows A1cs worsen in the teen years, not often improving until early adulthood (>25 years of age). While STePS has shown the rare capacity to move the needle on teens' glycemic control, a seemingly intractable outcome, it has not been tested in real-world contexts within existing pediatric diabetes programs.

Given the urgent need to translate research-based interventions into real-world settings, and the unacceptable lag-time between efficacy trials and routine uptake of clinical interventions, the investigators are currently conducting a type 1 hybrid effectiveness-implementation trial, funded by the ADA and by BreakthroughT1D (formerly known as Juvenile Diabetes Research Foundation), in 6 geographically distinct pediatric diabetes centers. Each center will enroll and randomly assign 60 economically, ethnically, and racially diverse teens aged 14-18 (N=360) to receive STePS either in-person (n=20) or via telehealth (n=20), or receive an educational telehealth control (n=20).

Design Considerations. The investigators will assess both effectiveness (primary outcomes) and implementation outcomes (secondary outcomes) via a Type 1 Hybrid Effectiveness Implementation design. The investigators chose a clinical effectiveness approach to evaluate STePS delivered in real-world contexts, using already-embedded behavioral health providers. The investigators prioritize external validity through recruiting a representative population, using an active comparison condition, and integrating the intervention into diabetes clinics. The investigators also chose an implementation approach to compare in-person versus telehealth strategies for improving uptake, fidelity, and sustainability of STePS. As noted by Curran et al. the time lag between research discovery and routine uptake is inflated by the step-wise progression of research from efficacy to effectiveness, and then only if effectiveness is established, to implementation. Blending effectiveness and implementation research is more desirable than pursing these lines of research independently and can "promote more rapid translational gains, more effective implementation strategies and more useful information for decision makers.

Effectiveness Outcomes: Improving Distress, A1c and Time-In-Range: Assessment of pre-post outcomes includes evaluating clinically meaningful changes in distress, A1c, and TIR. With respect to both A1c and TIR metrics, 0.3% is a clinically meaningful shift in the distribution of these measures of glycemic control as it generally represents about a 50% relative increase in the proportion of patients improving by 0.5% or more. However, 0.4% is generally accepted as evidence of a clinically meaningful change by the FDA. Therefore, if participant's A1c's improve by 0.4% at the end of 6 months, the investigators will conclude that STePS showed a clinically meaningfully improved metabolic control. With respect to diabetes-specific emotional distress, the minimal clinically important difference (MCID) of any psychosocial measure represents a threshold value of change in the score that represents a meaningful change in comparison to a statistically significant change. For this study, the investigators selected a stringent definition of MCID where the MCID is beyond the 95% confidence interval of the expected random variation in the distress score. For the PAID measures, that would be 8.3. Therefore, if participant's scores on the distress measures are reduced by >8.3 at the end of 6 months, then the study team will conclude that STePS has clinically meaningfully reduced distress. The investigators will also examine intervention delivery (in-person vs. telehealth) as a moderator of both STePS' effectiveness and implementation potential, increasing its potential for scalability.

Implementation Outcomes: The implementation approach is guided by two complementary frameworks: The Tailored Implementation in Chronic Diseases (TICD) framework, which supports the assessment of determinants (e.g., barriers and facilitators to chronic disease treatment ) that may impact STePS implementation in real-world diabetes clinics, and the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework, which guides an in-depth implementation evaluation, contrasting the two delivery approaches for STePS. The investigators will conduct a mixed-methods evaluation, collecting qualitative focus group data and implementation process data, contextualizing the effectiveness outcomes, and directly informing future efforts to bring STePS to scale. The investigators will conduct a mixed methods assessment of implementation outcomes. The original project only collects simple implementation data (e.g. acceptability, feasibility). The current proposal will conduct a significantly more robust and comprehensive implementation outcome evaluation. Data collection will include a series of surveys and focus group questions on the following domains: Reach will be captured by collecting data about: 1) recruitment (eligibility data); 2) enrollment (how many agreed/consented versus declined); 3) a demographic comparison of participants versus decliners, to assess representativeness of the participants. Adoption will be captured by assessing perceived barriers and facilitators of adopting STePS in real-world settings, determining if implementation of STePS is supportable in the pediatric diabetes clinics. Adoption will be assessed at the provider level via focus groups. At the provider level, the investigators will assess the opinions of the STePS interventionists, and of behavioral health providers who have diabetes-specific expertise, gathering opinions about adopting STePS in their centers. For both provider groups, the investigators will assess perceptions regarding the fit of STePS as a program that can be implemented in their clinical settings. Implementation will be captured via 1) feasibility of STePS implementation among interventionists and participants (e.g., interventionist training attendance, participant session attendance); 2) clinical trial feasibility data (retention and drop-out up rates); 3) perceived acceptability and appropriateness of STePS, reported by interventionists and participants, 4) fidelity to program delivery, with benchmarks including participants completing >80% of assigned homework and interventionists achieving >90% adherence to the treatment manual; and 5) costs associated with STePS implementation, both clinical implementation (e.g., provider hours spent training and delivering STePS) and research implementation costs (study team hours spent on recruitment, data collection, clinical supervision, etc.). Maintenance will assess perceived barriers and facilitators of the intervention's sustainability in pediatric diabetes clinics, allowing the investigators to understand how to best support STePS implementation, and guide future scale up efforts if STePS is proven to be effective.

Specific Aim 1. To test, in 336 teens across 6 clinical sites, the effectiveness of STePS in improving diabetes-specific emotional distress and preventing worsening glycemic control, both immediately post intervention and over time.

Hypothesis 1a: STePS will lead to clinically and statistically significant improvements in diabetes distress.

Hypothesis 1b: STePS will prevent the worsening of glycemic control (A1C and Time in Range) will not worsen over time. These hypotheses are consistent with the efficacy trial, and will prove effectiveness when implemented in real-world settings.

Specific Aim 2. To assess the implementation of STePS among key stakeholders (teen participants, interventionists). Recruitment, enrollment, representativeness, adoption, feasibility, acceptability, appropriateness, fidelity, costs and maintenance will be assessed as well as preferred implementation approaches.

Hypothesis 2a. Stakeholders will find few perceived barriers to implementing STePs and many perceived facilitators for adopting it in their clinical settings.

Hypothesis 2b. Implementation strategies will be plausible in diabetes clinics across the country.

The public health significance of these aims is strengthened by the focus on improving outcomes via a scalable, distress-reducing, resilience-building intervention.

ELIGIBILITY:
Inclusion Criteria: Eligibility criteria includes:

* T1D diagnosis for at least 1-year,
* using daily basal/bolus insulin,
* fluent in English,
* able to provide caregiver consent and teen assent to participate
* able to access telehealth via a digital device. We will focus recruitment on participants from populations under-represented in diabetes research (e.g., racial and ethnic minorities, families of low SES, using public aid, or living in rural communities).

Exclusion Criteria: To increase generalizability into typical clinical practice, exclusion criteria are minimal and include:

* cognitive or developmental disorders,
* participants cannot be a ward of the state.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2029-03-15 (Estimated); Study Completion 2029-03-15 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress | Distress is assessed at baseline, end of intervention (month 4.5), and then 6 (month 10.5) and 12 (month 16.5) months post intervention
  To assess clinically meaningful changes in DD, the minimal clinically important difference (MCID) represents a threshold value of change in the score that represents a meaningful change in comparison to a statistically significant change. For the PAID measures assessing distress we selected a stringent definition of MCID where the MCID is beyond the 95% confidence interval of the expected random variation in the distress score. For the PAID measures, that would be 8.3. Therefore, if participant's scores on the distress measures are reduced by >8.3 at the end of 6 months, then we will conclude that STePS has clinically meaningfully reduced distress.
Time in Range | Baseline, end of intervention (month 4.5) and again 6 (month 10.5) and 12 (month 16.5) months post intervention
  TIR is the percentage of time spent in the target glucose range of 70-180 mg/dL. Participants already using a continuous glucose monitor (CGM) will have their data downloaded at each of the 4 assessment time points. We will download data from the past 10 days at each assessment time-point, documenting percent time in range, percent time below 70 mg/dl and percent time above 180 mg/dL. For those not currently using a personal CGM we will give them a Dexcom Gen 6 Pro in a blinded fashion to use at each of the assessment time points. We are using blinded CGM for those without a personal CGM because data suggest that merely using a personal CGM can significantly improve TIR. Since giving participants a personal CGM with access to their data could in and of itself affect TIR, we have chosen to use blinded CGM for those participants so that we can collect the TIR range, but not negatively impact our ability to assess the TIR outcomes from participating in STePS.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Weissberg-Benchell, Ph.D., Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weissberg-Benchell J, Shapiro JB, Bryant FB, Hood KK. Supporting Teen Problem-Solving (STEPS) 3 year outcomes: Preventing diabetes-specific emotional distress and depressive symptoms in adolescents with type 1 diabetes. J Consult Clin Psychol. 2020 Nov;88(11):1019-1031. doi: 10.1037/ccp0000608. PMID 33136423
- See also: Study Website — https://www.luriechildrens.org/STEPST1D